CLINICAL TRIAL: NCT07088003
Title: Yoga as Mindful Movement: A Randomized Controlled Trial for Early Elementary School-Aged Children With Developmental Disabilities
Brief Title: Yoga as Mindful Movement: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Catherine Cook-Cottone, Professor, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBuffalo
Record Dates: First submitted 2025-07-11; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Developmental Disability
Keywords: Yoga; Mindfulness; Developmental Disability; Children; Early Elementary School
MeSH Terms: conditions — Developmental Disabilities | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga as Mindful Movement (Experimental)
  Interventions: Behavioral: Yoga as Mindful Movement
- Adapted Physical Education (Active Comparator)
  Interventions: Behavioral: Adapted Physical Education

INTERVENTIONS:
Behavioral: Yoga as Mindful Movement — YMM is an 8-week hybrid (in-person and virtual) school-based mindful yoga program (modified from its original 10-week, in-person design due to complications of COVID-19) informed by the teachings of Radiant Child Yoga. It was designed to teach students about self regulation through the integration of movement, breath, and present-moment awareness. It was delivered in the form of three, 30-minute YMM sessions each week by the same instructor-an individual with training and experience as an occupational therapist and yoga teacher through the Yoga Alliance and Radiant Child Yoga.
  Arms: Yoga as Mindful Movement
Behavioral: Adapted Physical Education — Adapted PE took place daily (Monday-Friday) for one hour and consisted of lessons on movement skills such as catching, throwing, aiming, running, jumping, skating, and dancing through various activities and games.
  Arms: Adapted Physical Education

SUMMARY:
This study aimed to close an existing research gap by exploring the impact of a school-based mindful yoga program, Yoga as Mindful Movement (YMM), on foundational motor skills, social-emotional competence, classroom behavior, attention, and impulse control of students with various developmental disabilities in kindergarten, first-, and second-grade (K-2).

ELIGIBILITY:
Inclusion Criteria: (a) Actively attending the participating school (indicating the presence of at least one developmental disability), (b) enrolled in kindergarten, first, or second grade, (c) part of a 6:1:3 classroom, (d) between the ages of 5 and 7, and (e) English-speaking

Exclusion Criteria: (a) Participant's family opted them out of the study, (b) participants was absent for three consecutive Yoga as Mindful Movement (YMM) classes

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Movement Assessment Battery for Children, Second Edition | From pre-enrollment (2 weeks before 8-week intervention) to post-enrollment (2 weeks after intervention's conclusion).
  The Movement Assessment Battery for Children, Second Edition measures children's motor performance in physical tasks (e.g., threading beads, catching a ball, walking heel-to-toe) through direct observation. Quantifiable criteria (e.g., task completion time, number of successful attempts, number of errors) is measured.
Devereux Student Strengths Assessment-Mini | From pre-enrollment (2 weeks before 8-week intervention) to post-enrollment (2 weeks after intervention's conclusion).
  This questionnaire asks assessors (classroom instructional staff) to rate how often a student displays certain behaviors (e.g., taking an active role in learning, making a suggestion or request in a polite way) in the past four weeks that correspond to social-emotional, cognitive, and interpersonal skills. Behaviors are rated on a 5-point Likert scale ranging from 0 (Never) to 4 (Very Frequently). A higher score indicates more social-emotional competence.
Child Behavior Rating Scale | From pre-enrollment (2 weeks before 8-week intervention) to post-enrollment (2 weeks after intervention's conclusion).
  The Child Behavior Rating Scale asks classroom instructional staff to indicate how often each student exhibits certain behaviors (e.g., returning to an unfinished task after interruption, attempting new challenging tasks) over the past week. This was completed using a 5-point Likert scale ranging from 1 (Never) to 5 (Always), with a higher score indicating positive behavior.
Head-Toes-Knees-Shoulders-Revised (HTKS-R) modified for Neurodiverse Learners (HTNL) | From pre-enrollment (2 weeks before 8-week intervention) to post-enrollment (2 weeks after intervention's conclusion).

SECONDARY OUTCOMES:
Classroom Observations | From enrollment to the end of treatment at 8 weeks
  Post-YMM (or adapted PE) session classroom observations of participants' behavior were conducted by two members of the research team who were masked to study conditions and not part of the school's instructional staff. Behaviors in nine categories (i.e., disrupting one's own or others' learning activity, demonstrating aggression toward staff or peers, engaging in a task, being prompted by an adult, affect, and wearing or not wearing a face mask-required due to COVID-19) were tracked and coded quantitatively. During each 30-minute observation block, three students per classroom were observed twice in 5-minute increments, for a total of 10 minutes each. This structure was implemented to capture potential variations in students' behavior over time. Because most classrooms had six students, the remaining three students were observed in the same manner the next time an observer visited the classroom.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine P. Cook-Cottone, PhD, Principal Investigator — University at Buffalo
Locations (1):
- Cantalician Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to concerns about participant privacy and limitations in the informed consent that prevent broader data sharing.